CLINICAL TRIAL: NCT01542957
Title: Cognitive Therapy for Unipolar Depression: Efficacy of a Dilemma-Focused Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: National Distance Education University (UNED) (Unknown); University of Minho (Other); University of Hertfordshire (Other); University of Bern (Other); University Ramon Llull (Other); Institut Trastorn Límit (Unknown); Hospital de Mataró (Other); Fundació Institut de Recerca de l (Unknown); Associació Centre de Salut Mental Nou Barris (Unknown); Fundacion IMIM (Other); EAP Poble Sec (Unknown); Associació Catalana de Terapies Cognitives (Unknown); Sant Pere Claver Fundació Sanitaria (Unknown)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dilemma2012; PSI2011-23246 (Other Grant/Funding Number: Ministry of Science and Innovation (Spanish Government))
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder
Keywords: Major Depressive Disorder; Dysthymic Disorder; Depression; Cognitive Behavior Therapy; Personal Construct Theory; Repertory Grid Technique; Cognitive Conflicts; Personal dilemmas
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral + Dilemma Therapy (Experimental): Combines Group Cognitive Behavioral Therapy with a Individual Dilemma-Focused Intervention
  Interventions: Behavioral: Combined Cognitive Behavioral and Dilemma-Focused Therapy
- Cognitive Behavioral Therapy (Active Comparator): Combined Group and Individual Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy for Depression

INTERVENTIONS:
Behavioral: Combined Cognitive Behavioral and Dilemma-Focused Therapy — 7 2-hour sessions of Group Cognitive Behavioral Therapy for Depression + 8 individual sessions of a Dilemma-Focused Intervention + 1 3-hour final group session. Manualized.
  Other Names: Personal Construct Therapy
  Arms: Cognitive Behavioral + Dilemma Therapy
Behavioral: Cognitive Behavioral Therapy for Depression — Cognitive Behavioral Therapy for Depression. Format: 7 2-hour sessions in group + 8 individual sessions + 1 3-hour final group session. Manualized.
  Other Names: Cognitive Therapy
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to determine the efficacy of a brief psychological intervention focused on the personal dilemmas identified for each depressive patient. For that, this intervention is combined to group cognitive therapy (an already proven efficacious format) and compared to cognitive individual therapy.

DETAILED DESCRIPTION:
Depression is one of the more severe and serious health problems because of its morbidity, disabling effects and for its societal and economic burden. Despite the variety of existing pharmacological and psychological treatments most of the cases evolve with only partial remission, relapse and recurrence.

Cognitive models made a significant contribution in the understanding of unipolar depression and its psychological treatment. Even though, success is only partial and many authors affirm the need to improve those models and also the treatment programs derived from them. One of the issues that requires further elaboration is the difficulty these patients experience in responding to treatment and in maintaining therapeutic gains across time without relapse or recurrence.

Our research group has been working in the notion of cognitive conflict viewed as personal dilemma according to personal construct theory. The investigators use a novel method for identifying those conflicts using the repertory grid technique. Preliminary results with depressive patients show that more than 90% of them have one or more of those conflicts. This fact might explain the blockage and the difficult progress of these patients, especially the more severe and/or chronic. These results justify the need for specific interventions focused in the resolution of these internal conflicts.

This study aims to empirically test the hypothesis that an intervention focused on the dilemma(s) specifically detected for each patient will contribute to enhance the efficacy of Cognitive-Behavioral Therapy for depression. A therapy manual for this approach will be tested using a randomized clinical trial by comparing the outcome of two treatment conditions: a CBT treatment package and another package combining cognitive-behavioral and dilemma-focused interventions. The investigators expect that this combined package will increase the efficacy of CBT, one of the more prestigious therapies for depression, this resulting in a significant contribution for its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meeting diagnostic criteria for Major Depressive Disorder (MDD) or Dysthymic Disorder (DD) according to the DSM-IV-TR (APA, 2002) criteria a assessed using SCID-I
* A score above 19 on the BDI-II Questionnaire
* Presenting at leat one cognitive conflict (implicative dilemma or dilemmatic construct) as assessed using the Repertory Grid Technique
* Enough level of competence to communicate in Spanish or Catalan

Exclusion Criteria:

* Bipolar disorders
* Psychotic symptoms
* Substance abuse
* Organic brain dysfunction
* Mental retardation
* Serious suicidal ideation
* Receiving psychological treatment (unless it is suspended at the time of inclusion in the study itself, in agreement with the patient and the practitioner applying it)
* Substantial visual, hearing or cognitive deficits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, Ph.D., Principal Investigator — University of Barcelona
Locations (4):
- Spain (4):
  - Hospital de Mataro (Consorci Sanitari del Maresme), Mataró, Barcelona
  - CAP Les Hortes, Barcelona, Catalonia
  - Fundació Sanitària Sant Pere Claver, Barcelona, Catalonia
  - Associació Catalana de Teràpies Cognitives, Barcelona, Catalonia

REFERENCES:
- [Background] Feixas G, Bados A, Garcia-Grau E, Montesano A, Dada G, Compan V, Aguilera M, Salla M, Soldevilla JM, Trujillo A, Paz C, Botella L, Corbella S, Saul-Gutierrez LA, Canete J, Gasol M, Ibarra M, Medeiros-Ferreira L, Soriano J, Ribeiro E, Caspar F, Winter D. Efficacy of a dilemma-focused intervention for unipolar depression: study protocol for a multicenter randomized controlled trial. Trials. 2013 May 17;14:144. doi: 10.1186/1745-6215-14-144. PMID 23683841
- [Result] Feixas G, Bados A, Garcia-Grau E, Paz C, Montesano A, Compan V, Salla M, Aguilera M, Trujillo A, Canete J, Medeiros-Ferreira L, Soriano J, Ibarra M, Medina JC, Ortiz E, Lana F. A DILEMMA-FOCUSED INTERVENTION FOR DEPRESSION: A MULTICENTER, RANDOMIZED CONTROLLED TRIAL WITH A 3-MONTH FOLLOW-UP. Depress Anxiety. 2016 Sep;33(9):862-9. doi: 10.1002/da.22510. Epub 2016 Apr 22. PMID 27103215
- [Derived] Feixas G, Paz C, Garcia-Grau E, Montesano A, Medina JC, Bados A, Trujillo A, Ortiz E, Compan V, Salla M, Aguilera M, Guasch V, Codina J, Winter DA. One-year follow-up of a randomized trial with a dilemma-focused intervention for depression: Exploring an alternative to problem-oriented strategies. PLoS One. 2018 Dec 13;13(12):e0208245. doi: 10.1371/journal.pone.0208245. eCollection 2018. PMID 30543642
- See also: Web page in Spanish and Catalan describing the research project and recruitment information — http://www.ub.edu/terdep

RESULTS

PARTICIPANT FLOW:
Period: End of Therapy
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Started | 65 | 63
Completed | 53 | 53
Not Completed | 12 | 10
Period: 3-month Follow-up
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Started | 53 | 53
Completed | 50 | 45
Not Completed | 3 | 8
Period: 12-month Follow-up
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Started | 53 | 53
Completed | 37 | 40
Not Completed | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.37 (11.22) | 50.06 (11.03) | 49.20 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 99
  Male | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Beck Depression Inventory-Second Edition (BDI-II) at the End of Therapy, 3 and 12-month Follow-up
Description: To assess change in severity of depressive symptoms. The Total score is reported, which is the sum of the ratings of all items and ranges from 0 to 63, with higher scores indicating more severity of depressive symptoms.
Time Frame: End of therapy (16 weeks), 3 and 12-month follow-up
Population: The overall number of participants analyzed are those who completed the treatment but not all of them completed follow-up assessments at 3 and 12-month after the end of the therapy. In each row the number of those participants who completed the assessment are specified
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 53 | 53
units on a scale
  Baseline | 37.23 (8.96) | 36.94 (9.56)
  At the end of therapy change from baseline | -17.62 (12.05) | -15.52 (13.92)
  3-month follow-up change from baseline: number analyzed (Participants) | 50 | 45
  3-month follow-up change from baseline | -15.42 (13.16) | -15.60 (15.56)
  12-month follow-up change from baseline: number analyzed (Participants) | 37 | 40
  12-month follow-up change from baseline | -19.51 (13.17) | -16.65 (13.87)
Statistical Analysis 1: Comparison: Cognitive Behavioral + Dilemma Therapy vs Cognitive Behavioral Therapy; Test type: Superiority or Other; p = 0.60, Mixed Models Analysis; Slope = -0.96, 95% CI 2-sided [-3.35 to 1.43], Standard Error of Mean 0.69

2. Secondary Outcome: Change From Baseline in Hamilton-Depression Rating Scale-17 Items
Description: This clinician-administered measure was only applied to 78 patients at pre- and posttreatment. It measures severity of depressive symptoms. The Total score is reported, which is the sum of the ratings of all items and ranges from 0 to 54, with higher scores indicating more severity of depressive symptoms.
Time Frame: End of therapy and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 42 | 38
units on a scale
  Baseline | 18.93 (6.96) | 20.05 (6.09)
  At the end of therapy change from baseline | -7.61 (9.21) | -8.84 (8.28)
  12 month follow-up change from baseline: number analyzed (Participants) | 31 | 28
  12 month follow-up change from baseline | -5.32 (9.56) | -7.89 (9.57)
Statistical Analysis 1: Comparison: Cognitive Behavioral + Dilemma Therapy vs Cognitive Behavioral Therapy; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis; Slope = 1.27, 95% CI 2-sided [-0.71 to 3.25], Standard Error of Mean .53

3. Secondary Outcome: Change From Baseline in Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) at the End of Therapy, 3 and12 Month Follow-up
Description: To assess subjective well-being, symptoms or problems, life functioning, and risk. The Total score is reported, which is the sum of the ratings of all items divided by the number of items (34). The score and ranges from 0 to 4, with higher scores indicating more severity of psychological distress.
Time Frame: End of therapy, 3 and 12 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 53 | 53
units on a scale
  Baseline | 2.17 (0.50) | 2.08 (0.56)
  At the end of therapy change from baselina | -0.76 (0.70) | -0.67 (0.75)
  3 month follow-up change from baseline: number analyzed (Participants) | 50 | 45
  3 month follow-up change from baseline | -0.59 (0.76) | -0.63 (0.80)
  12 month follow-up change from baseline: number analyzed (Participants) | 37 | 40
  12 month follow-up change from baseline | -0.77 (0.81) | -0.58 (0.86)
Statistical Analysis 1: Comparison: Cognitive Behavioral + Dilemma Therapy vs Cognitive Behavioral Therapy; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis; Slope = -0.01, 95% CI 2-sided [-0.14 to 0.12]

ADVERSE EVENTS:
Description: "0" means that serious and other [non-serious] adverse events were not collected or assessed as part of the study since no detrimental effects were expected as result of psychotherapies.
Arm/Group | Cognitive Behavioral + Dilemma Therapy | Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes